CLINICAL TRIAL: NCT00014729
Title: Phase I Study of Isotretinoin in Patients With Recessive Dystrophic Epidermolysis Bullosa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/15738; UNCCH-FDR001796
Record Dates: First submitted 2001-04-10; First posted 2001-04-11 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-05

CONDITIONS: Epidermolysis Bullosa
Keywords: dermatologic disorders; epidermolysis bullosa; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Epidermolysis Bullosa; Skin Diseases; Genetic Diseases, Inborn; Rare Diseases | interventions — Isotretinoin

INTERVENTIONS:
Drug: isotretinoin

SUMMARY:
OBJECTIVES:

I. Determine the safety of isotretinoin in patients with recessive dystrophic epidermolysis bullosa.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients receive oral isotretinoin daily for 8 months in the absence of disease progression or unacceptable toxicity.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of recessive dystrophic epidermolysis bullosa (RDEB) RDEB Hallopeau-Siemens OR RDEB non-Hallopeau-Siemens
* Concurrent enrollment in the National Epidermolysis Bullosa Registry
* No regional or distant metastasis in patients with previous or concurrent squamous cell carcinoma

--Patient Characteristics--

* Hepatic: No clinically significant hypertriglyceridemia No clinically significant hepatic dysfunction
* Renal: No clinically significant renal dysfunction
* Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2000-10; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Jo-David Fine, Study Chair — University of North Carolina